CLINICAL TRIAL: NCT03611439
Title: Effects of an 8 Component Botanical Supplement on Mild and Moderate Alzheimer's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genescient Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Genescient
Record Dates: First submitted 2018-07-17; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Alzheimer Disease; Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, double blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReBuilder Actives (Active Comparator): Subjects take one 650 mg capsule by mouth twice a day for 12 months.
  Interventions: Dietary Supplement: ReBuilder
- ReBuilder Placebo (Placebo Comparator): Subjects take one placebo capsule by mouth twice a day for 12 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ReBuilder — 8-component botanical dietary supplement
  Other Names: MX100A; Memex+
  Arms: ReBuilder Actives
Dietary Supplement: Placebo — Inactive Placebo Capsule
  Arms: ReBuilder Placebo

SUMMARY:
This placebo-controlled, double blind study evaluates the treatment effects of adding a multi-pathway botanical dietary supplement (ReBuilder) to the standard treatment regimens of subjects diagnosed with mild or moderate stage Alzheimer's Disease. The objective of the study is to determine if mild and moderate AD patients exhibit improved or stabilized cognitive function when this supplement is added to maximum tolerated doses of their standard treatments.

DETAILED DESCRIPTION:
Currently, there is no treatment that can stop the progression of Alzheimer's Disease. The investigators in this study have used transgenic Drosophila melanogaster models and machine learning to develop an eight component botanical mixture (Geneaire™* ReBuilder™) that targets multiple genetic pathways involved in brain aging and dementia that are homologous between Drosophila and humans.

While beta-amyloid plaques and phosphorylated-tau tangles are diagnostic for AD, the cause(s) of their soluble precursors that kill neurons has not been determined. The majority of AD patients are diagnosed after 60 years of age. Many studies point to aging related processes like inflammation, neural vascular damage, neural stress, altered cell metabolism, inefficient cellular autophagy, microglial dysfunction, mitochondrial dysfunction, and poor diet as potential causal factors in the decline of brain function over the decades that precede an actual AD diagnosis. AD is a multifaceted pathology involving many biochemical pathways and thus a multifaceted therapeutic approach may prove beneficial.

The goal of this study was to test ReBuilder on human cognitive function. During the 12-month pilot study, the subjects were evaluated quarterly on the Mini Mental State Exam (MMSE), Alzheimer's Disease Cooperative Study's Activities of Daily Living (ADCS-ADL), and the Clinical Dementia Rating Sum of Boxes (CDR-SB).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed mild or moderate Alzheimer's Disease

Exclusion Criteria:

* History of heart disease
* History of heart attack
* History of cancer
* History of stroke or transient ischemic attack

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-12-25 (Actual); Study Completion 2015-12-25 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Mini Mental State Exam (MMSE) Scores | Change from baseline MMSE at 12 months
  dementia questionnaire
Change From Baseline Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Scores | Change from baseline ADCS-ADL at 12 months
  daily living activity questionnaire
Change From Baseline Clinical Dementia Rating Sum of Boxes (CDR-SB) Scores | Change from baseline CDR-SB at 12 months
  dementia assessment